CLINICAL TRIAL: NCT06996041
Title: Effect of Chocking First Aid Management Program on Knowledge, Attitude and Practice of Health Care Support Workers.
Brief Title: Chocking First Aid Management Program for Health Care Support Workers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rec/ 02048 Tanveer Kakar
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Choking
Keywords: Knowledge; Attitude; Practice; Chocking first aid
MeSH Terms: conditions — Airway Obstruction; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chocking first aid management program (Experimental): Power point presentation , Video demonstration, and Practical demonstration of chocking first aid management
  Interventions: Other: Chocking first aid management program

INTERVENTIONS:
Other: Chocking first aid management program — Power point presentation , Video demonstration, and Practical demonstration of chocking first aid management

SUMMARY:
To determine the effect of chocking first aid awareness program on knowledge, attitude and practice of health care support workers. Despite the importance of first aid skills, there may be gaps in the knowledge of healthcare support workers regarding choking management. A well-designed program can address these gaps, ensuring that workers are aware of the latest guidelines and techniques for managing choking incidents.

Knowledge and attitudes alone are not sufficient; practical skills are crucial. The program aims to translate theoretical knowledge and positive attitudes into effective practice. Training can enhance the workers' ability to perform first aid procedures correctly and confidently.

DETAILED DESCRIPTION:
It is very important for every person in the community to know about first aid training to save lives and improve the overall quality of community health. Health care professionals and trainees are expected to know about it, as they frequently face life threatening situations in their daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Physical Therapist
* Pharmacists
* Lab Technicians
* Minimum 1 Year of Practice

Exclusion Criteria:

* Unwilling
* Any upper-limb MSK problem
* Recent certification on emergency management

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge, Attitude and Practice of Chocking first aid | 2 weeks
  Changes from baseline to post-intervention program, assessed through KAP Questionnaire with three parts, Questions to assess first aid choking knowledge, attitude towards choking first aid and practice on choking first aid. Highest score shows good knowledge , positive attitude and good practice.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MS-CPPT PhD*, Principal Investigator — Riphah International University
Locations (1):
- Northwest General Hospital & Research Center and Northwest Institute Of Health Sciences, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No